CLINICAL TRIAL: NCT06759883
Title: Local Dishes Versus Ready-to-use Therapeutic Foods in the Management of Severe Acute Malnutrition During the Rehabilitation Phase: a Randomized, Single-blind Study at the Regional Hospital Annex of Mokolo (Cameroon)
Brief Title: Local Dishes Versus Ready-to-use Therapeutic Foods Management of Severe Acute Malnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Garoua (Other)
Responsible Party: Principal Investigator, KAMO SELANGAI Hélène, Principal Investigator, University of Garoua
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 062/24L/MSP/DRSP-EN/HRA-MOK
Record Dates: First submitted 2024-12-15; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Effect of Food; Malnourished Children
Keywords: Efficacy; Local dishes; Severe acute malnutrition; Rehabilitation phase
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind study
Who Masked: Participant
Masking Description: Participants were assigned an order number based on their arrival. Those with an even number were placed in the control group (under ECDT) following the national protocol, while those with an odd number were placed in the experimental group (using local dishes with nutritional education).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ready-to-use therapeutic foods (No Intervention): Control group on ready-to-use therapeutic foods
- Local Dishes (Experimental): Intervention group with local dishes
  Interventions: Combination Product: local dishes using the my plate concept

INTERVENTIONS:
Combination Product: local dishes using the my plate concept — The intervention in this study consists of replacing the ready-to-use therapeutic foods prescribed in phase 2 of the management of acute severe malnutrition with balanced local dishes.
  Other Names: well-balanced local dishes
  Arms: Local Dishes

SUMMARY:
In a context of frequent shortages of ready-to-use therapeutic foods (RUTFs), this study aimed at assessing the effectiveness of the use of local dishes in conjunction with nutritional education for children with severe acute malnutrition (SAM) during the rehabilitation phase. This work is based on a randomized, single-blind study. Children aged between 6 to 59 months, hospitalized for SAM and undergoing treatment during the rehabilitation phase, were included. Randomization was performed by consecutive inclusion based on:

* Even numbers (control group under RUTFS) and
* Odd numbers (intervention group with local dishes).

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effectiveness of using local dishes combined with nutritional education in children with severe acute malnutrition (SAM) during the rehabilitation phase. Specifically, the aim was to compare the evolution of clinical parameters (weight, mid-upper arm circumference, length of hospital stay) during treatment, determine the effectiveness of using local dishes combined with nutritional education in the management of SAM, and assess the outcomes of the treated children. This was a randomized, single-blind study conducted over an 11-month period spanning from October 2023 to June 2024 at the In house therapeutic nutrition centre (ITNC) of the Mokolo Regional hospital Annex in the Far North region of Cameroon. The population undergoing the study consisted of children aged between 6 to 59 months hospitalized in the ITNC ward for severe acute malnutrition in the rehabilitation phase. The sample size was calculated using Kelsey's formula.

The minimum sample size required was 24 All patients aged between 6 and 59 months with severe acute malnutrition undergoing treatment in the rehabilitation phase, whose parents or guardians had provided consent by signing the consent form, were included. Patients suffering from identified chronic conditions such as tuberculosis, heart disease, etc., were excluded. Patient recruitment was conducted in collaboration with community workers, who facilitated communication with parents or guardians.

During the procedure, discussion sessions were held, focusing primarily on malnutrition awareness, food groups, child weaning, and practical cooking workshops with the parents. Randomization was conducted using the consecutive allocation method based on even and odd numbers. Participants were assigned an order number based on their arrival. Those with an even number were placed in the control group following the national protocol, while those with an odd number were placed in the experimental group (using local dishes with nutritional education).

The meals consisted of a variety of local dishes. Mothers selected menus typically consumed in their homes, prepared them under usual conditions, and then fed their children the quantities accepted by the child. The interviewer ensured that each meal was balanced and included the five food groups of the "My Plate" concept.

The follow-up of selected patients was divided into a hospital phase lasting 3 days and a community phase, with daily follow-ups conducted at regular intervals.

Data collected was recorded on a survey form. For the child's physical examination, the investigator used WHO Z-score curves, vital sign monitoring equipment, a electronic scale ,a UNICEF infant meter, and a paediatric MUAC tape measure from UNICEF.

The survey form collected data on:

Socio-demographic characteristics of the parents or guardians of the children. Clinical and nutritional characteristics: child's age, sex, breastfeeding method, type of malnutrition, vaccination status, Z-score at admission, mid-upper arm circumference (MUAC) at admission and discharge, duration of the rehabilitation phase, medical complications, and Z-score at discharge.

Monitoring and progress during treatment: vital parameters (temperature, heart rate, pulse), anthropometric data (weight, height, Z-score, blood pressure), clinical parameters, and weight progression.

Therapeutic outcomes: cured, relapse, or death. The data collected were analysed using IBM SPSS 27 and organized in Microsoft Office Excel 2019. Statistics tests used were the chi-square test, Fisher's exact test, and Student's t-test. Categorical variables were described as percentages, proportions, and/or frequencies. For statistical analyses, an α error threshold of 5% was applied, and means were expressed with 95% confidence intervals. P-values < 0.050 were considered statistically significant.

The research protocol was submitted to the regional ethics committee and received approval under ethics clearance number 0065/CERH/NO/2024. Parental consent was obtained prior to inclusion. No invasive procedures were performed, and parents were free to decline participation without any impact on their child's follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged between 6 and 59 months
* with severe acute malnutrition undergoing treatment in the rehabilitation phase,
* whose parents or guardians had provided consent by signing the consent form,

Exclusion Criteria:

* Patients suffering from identified chronic conditions such as HIV/AIDS, tuberculosis, heart disease,

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Correlation between the number of grams (g) of weight gain and the treatment option used | From enrolment to the end of treatment up to 12 Weeks
  Describe the difference observed between the control and intervention groups in terms of weight gain at the end of hospitalization.

SECONDARY OUTCOMES:
Correlation between number of hospital days (days) and therapeutic option used | From enrolment to the end of treatment up to 12 Weeks
  Describe the difference observed between the control and intervention groups in terms of the number of days spent in hospital.

OTHER OUTCOMES:
Correlation between patient outcome relapse and treatment option used in both groups at the end of the study. | From enrolment to the end of treatment up to 12 Weeks
  Describe the outcome of participants in the two study groups With regard to relapse
Correlation between patient outcome deaths and treatment option used in both groups at the end of the study. | From enrolment to the end of treatment up to 12 Weeks
  Describe the outcome of participants in the two study groups With regard to deaths

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Sap, Pediatrician, Study Director — Faculty of Medicine and Biomedical Sciences University of University of Yaoundé
Locations (1):
- Faculty of Medicine and Biomedical Science, Garoua, North Region, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared in the form of a publication in a paediatric journal
Supporting Information: SAP, ICF
Time Frame: Unending Beginning 6month after publication
Access Criteria: After publication

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT06759883/SAP_000.pdf
  • Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT06759883/ICF_001.pdf